CLINICAL TRIAL: NCT00793520
Title: Effect of Milnacipran on Pain Processing and Functional Magnetic Resonance Imaging (fMRI) Activation Patterns in Patients With Fibromyalgia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: James Perhach, PhD, Executive Director, Clinical Development, Neurology, Forest Research Insititute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MLN-MD-16
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Results first posted 2010-07-01 (Estimated); Last update posted 2010-07-01 (Estimated); Status verified 2010-06

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; milnacipran; Forest Laboratories
MeSH Terms: conditions — Fibromyalgia | interventions — Milnacipran

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Twice daily oral administration of milnacipran for 5 weeks, placebo for 2 weeks, and crossover to placebo for 5 weeks.
  Interventions: Drug: Milnacipran; Drug: Placebo
- 2 (Experimental): Twice daily oral administration of placebo for 5 weeks, placebo for 2 weeks, and crossover to milnacipran for 5 weeks.
  Interventions: Drug: Placebo; Drug: Milnacipran

INTERVENTIONS:
Drug: Milnacipran — Twice daily oral administration of Milnacipran for 5 weeks.
  Arms: 1
Drug: Placebo — Twice daily oral administration of placebo for 5 weeks.
  Arms: 2
Drug: Placebo — Twice daily oral administration of placebo for 5 weeks.
  Arms: 1
Drug: Milnacipran — Twice daily oral administration of Milnacipran for 5 weeks.
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the effect of milnacipran on how the brain processes pain in patients with fibromyalgia and to assess the relationship between this effect and brain activation patterns during functional magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of fibromyalgia defined by 1990 American College of Rheumatology (ACR) criteria
* Visual analog pain score between 40 and 90 mm
* Right-hand dominance

Exclusion Criteria:

* Suicidal risk
* Substance Abuse
* Pulmonary dysfunction
* Renal impairment
* Active cardiac disease
* Autoimmune disease
* Uncontrolled narrow-angle glaucoma
* Active liver disease
* Cancer
* Active peptic ulcer disease or a history of inflammatory bowel disease or celiac sprue
* Unstable endocrine disease
* Prostatic enlargement

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-11; Primary Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allan Spera, Study Director — Forest Research Institute, a subsidiary of Forest Laboratories Inc
Locations (1):
- Forest Investigative Site, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from November 2008 to April 2009 at one university location.
Pre-assignment Details: Of the five enrolled patients, only two received double-blind study medication due to equipment failure at the study site.
Groups:
- Milnacipran to Placebo: Twice daily oral administration of milnacipran for 5 weeks, placebo for 2 weeks, and crossover to placebo for 5 weeks.
- Placebo to Placebo: Twice daily oral administration of placebo for 5 weeks, placebo for 2 weeks, and crossover to milnacipran for 5 weeks.
Period: Milnacipran Crossover to Placebo
Arm/Group | Milnacipran to Placebo | Placebo to Placebo
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Period: Placebo Crossover to Milnacipran
Arm/Group | Milnacipran to Placebo | Placebo to Placebo
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Milnacipran to Placebo | Placebo to Placebo | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 37 | 48 | 42.5 (7.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Secondary Outcome: Change in Diffuse Noxious Inhibitory Control (DNIC) Effect From Baseline to End of Treatment.
Description: DNIC is evaluated using a conditioning stimulus and a test stimulus. Painful blunt pressure is applied to the thumbnail of the patient's left hand for 30 sec. Patient rates pain experienced on numerical scale of 0(no pain) to 100(worst pain) at 10, 20 & 30 sec. This is repeated 3 times and a mean pain score is calculated. 5 minutes following test stimulus, patient's right hand is immersed in 12C water at 30 sec test stimulus is reapplied and a 2nd mean pain score is calculated. The difference in mean pain rating before and after conditioning stimulus indicates presence and magnitude of DNIC
Time Frame: Weeks 0, 5, 7 and 12
Measure: Mean (95% Confidence Interval); unit: Pain Rating
Arm/Group | Milnacipran to Placebo | Placebo to Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change in Medium Pressure Pain Threshold From Baseline to End of Treatment.
Description: Pain intensity is rated using the Gracely Box Scale, where 0 is no pain sensation and 20 is extremely intense. Painful blunt pressure is applied to the thumbnail of the patient's left hand. A software system will determine medium(rated as 7 or 8) and high pain (rated as 13 or 14) thresholds at baseline, week 5 and at a second baseline at week 7 and week 12.
Time Frame: Week 0, 5, 7 and 12
Measure: Mean (95% Confidence Interval); unit: Kg
Arm/Group | Milnacipran to Placebo | Placebo to Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Milnacipran: Twice daily oral administration of milnacipran for 5 weeks, placebo for 2 weeks, and crossover to placebo for 5 weeks.
- Placebo: Twice daily oral administration of placebo for 5 weeks, placebo for 2 weeks, and crossover to milnacipran for 5 weeks.
Arm/Group | Milnacipran | Placebo
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Milnacipran (N=1) | Placebo (N=1)
Food poisoning (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Nightmares (Psychiatric disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects enrolled. Technical problems with MRI equipment resulted in early study termination. No analysis was performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No